CLINICAL TRIAL: NCT00647829
Title: Clinical Protocol For A Double-Blind, Randomized, Placebo-Controlled Comparison Of The Efficacy, Safety, And Tolerability Of Bextra® (Valdecoxib) 20 Mg Twice Daily, Bextra® 40 Mg Once Daily, And Placebo In The Symptomatic Treatment Of Subjects With Pharyngitis
Brief Title: A Comparison Of Valdecoxib 20 Mg Twice Daily and 40 Mg Daily and Placebo In The Treatment Of Sore Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3471026
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Pharyngitis
Keywords: pharyngitis, sore throat
MeSH Terms: conditions — Pharyngitis | interventions — valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 20 mg tablet by mouth twice daily (BID) for 2 doses over a 24-hour period
  Arms: Arm 1
Drug: valdecoxib — valdecoxib 40 mg tablet by mouth once daily (QD) for 2 doses over a 24-hour period
  Arms: Arm 2
Drug: placebo — placebo tablet by mouth for 2 doses over a 24-hour period
  Arms: Arm 3

SUMMARY:
The study was performed to evaluate the analgesic efficacy, safety, and tolerability of valdecoxib 20 mg twice daily (BID), valdecoxib 40 mg once daily (QD), and placebo in patients with moderately to severely painful symptomatic sore throat over a 24-hour period. In addition, the study was to validate a new scale and criteria for measuring pain in sore throat and evaluate the effects of selective serotonin reuptake inhibitors and past sore throat pain on pain score and efficacy of analgesics. The study also examined what type of medications are commonly used for sore throat and whether this information has relevance to analgesic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Included patients had moderate to severe pain, as measured by the Sore Throat Pain Intensity Scale (STPIS) on swallowing ≥66 mm on a 100-mm visual analogue scale (VAS) and a minimum of 4 points on the 10-point Tonsillo-Pharyngitis Score (TPS) but who were not coughing or experiencing any evidence of mouth-breathing.

Exclusion Criteria:

* Patients who used throat lozenges, throat spray, cough drops or menthol-containing products within 2 hours, short-acting analgesics/antipyretics (eg, ibuprofen) or any form of cold medication within 8 hours, antibiotics for acute disease within 24 hours of first dose of study medication, or presumed diagnosis of infectious mononucleosis, known allergy or hypersensitivity to NSAIDs, COX-2 specific inhibitors, sulfonamides, or acetaminophen were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2003-02; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Sum of Sore Throat Pain Intensity Difference (SPID, VAS) on swallowing | 2-hour period after the first dose

SECONDARY OUTCOMES:
Sum of Sore Throat Pain Intensity Difference (SPID, VAS) on swallowing | 4, 6, 8, 10, 12, and 24 hours after first dose
Peak Sore Throat Pain Intensity Difference (PPID) on swallowing | 24-hour period after the first dose
Throat Soreness Difference (TSD) on swallowing | each post dose time point
Sum of Throat Soreness Difference (STSD) on swallowing | 2, 4, 6, 8, 10, 12, and 24 hours after first dose
Peak Throat Soreness Difference (PTSD) on swallowing | 24-hour period after the first dose
Sum of Sore Throat Relief Rating (SSTRR) on swallowing | 2, 4, 6, 8, 10, 12, and 24 hours after first dose
Peak Sore Throat Relief Rating (PSTRR) on swallowing | 24-hour period after the first dose
Time to onset of analgesia | 2-hour period after the first dose
Time to rescue medication | 24-hour period after the first dose
Patient's global evaluation of study medication | 24-hour period after the first dose
Percent of patients taking rescue medications | 24-hour period after the first dose
Sore Throat Relief Rating (STRR) on swallowing | post dose time point
Patient's satisfaction with treatment | 24-hour period after the first dose
Sore Throat Pain Intensity Difference (PID, VAS) on swallowing | each post dose time point
Time to perceptible pain relief | 2-hour period after the first dose
Time to meaningful pain relief | 2-hour period after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Storrs, Connecticut
  - Pfizer Investigational Site, Boca Raton, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3471026&StudyName=Double-Blind%2C%20Randomized%20Protocol%20For%20Comparison%20Of%20The%20Efficacy%2C%20And%20Safety%20Of%20Valdecoxib%2020%20Mg%20Twice%20Daily%2C%20Valdecoxib%2040%20Mg%20Dai